CLINICAL TRIAL: NCT04348604
Title: Improving Adherence in Adolescents and Young Adults With Bipolar Disorder
Acronym: IGNITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH117206 (NIH)
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized Adherence Enhancement for AYA (Experimental): This arm will receive the experimental intervention, Customized Adherence Enhancement for Adolescents and Young Adults (CAE-AYA).
  Interventions: Behavioral: Customized Adherence Enhancement for Adolescents and Young Adults (CAE-AYA)
- Enhanced Treatment as Usual (ETAU) (Active Comparator): This arm will receive the control intervention, Enhanced Treatment as Usual (ETAU).
  Interventions: Behavioral: Enhanced Treatment as Usual (ETAU)

INTERVENTIONS:
Behavioral: Customized Adherence Enhancement for Adolescents and Young Adults (CAE-AYA) — Customized Adherence Enhancement for Adolescents and Young Adults (CAE-AYA): CAE-AYA participants will have 4 core in-person sessions (45-60 minutes each) spaced about 1 week apart over a period of approximately 4 weeks and one "booster" in-person session approximately 4 weeks after completion of the 4 core sessions (total of up to 5 in-person sessions spaced out over 8 weeks). There will be one follow-up phone call with a study interventionist, approximately 6 weeks post-baseline (timed half-way between completion of the core sessions and the "booster" session). All AYAs assigned to the CAE-AYA arm will receive all 4 modules (Psychoeducation on BD Medications; Communication with Providers & Caregivers; Medication Routines; and Targeting Risky Behavior via Modified Motivational Enhancement Therapy (MET)), with the content within each module being customized to developmental stage and behavioral experience.
  Arms: Customized Adherence Enhancement for AYA
Behavioral: Enhanced Treatment as Usual (ETAU) — Enhanced Treatment as Usual (ETAU): ETAU will consist of usual clinical care with prescribing clinicians and therapists, augmented by written materials specific to BD for AYAs and 6 follow-up telephone calls to briefly review the materials and be available for questions by social workers with mental health experience and at least some experience in working with AYA with BD. In order to ensure that there is not treatment contamination, different trained interventionists will be used for CAE and eTAU. Therapists will briefly review the materials and be available for questions during the phone calls. Materials will cover general self-management in BD. The calls will be relatively brief (maximum of 20-30 minutes).
  Arms: Enhanced Treatment as Usual (ETAU)

SUMMARY:
Although poor medication adherence occurs in more than 65% of adolescent and young adults (AYA) with bipolar disorder (BD) and is associated with poor recovery, high rates of relapse, and a 5.2 fold increased suicide risk, there have been no interventions that specifically target adherence in AYA with BD. This proposal will modify and test a customized adherence enhancement (CAE) intervention developed by the investigative team and found to be effective in BD adults in a high-risk, high-need group: AYAs with BD who are poorly adherent with prescribed BD medications. The project addresses the critical need for evidence-based interventions to improve adherence in AYAs with BD and has the potential to change outcome trajectories in high-risk young people with BD as they transition to adulthood.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of bipolar disorder (BD), type I or II as diagnosed by the Structured Clinical Interview for DSM-5 (SCID-5)
* Poor adherence defined as missing ≥ 20% of prescribed evidence-based BD medications, i.e., mood stabilizer (e.g., lithium, valproic acid, or carbamazepine) or second generation antipsychotics, on the TRQ for the past week or past month
* If < 18 years, able and willing to give written informed assent and have a legal guardian provide written informed consent; if > 18 years, able and willing to provide written informed consent
* Fluent in English

Exclusion Criteria:

* Unable to receive care in the outpatient setting due to illness severity
* A DSM-5 diagnosis of an autism spectrum disorder or primary psychotic disorder
* Documented or suspected IQ < 70
* Prior enrollment in CAE or Phase 2
* Have recently (in the past month) started a new psychotherapy/behavioral intervention

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Universty, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data entered into the NIMH National Database: We will collaborate with our project office to determine the best mechanism to ensure that our Phase 3 data is entered into the common informatics platform by NIMH, called the National Database for Clinical Trials Related to Mental Illness (http://ndct.nimh.nih.gov, NDCT). We will work with NIMH to transform the data we collect into relevant information using the suggested consent form language, NIMH software that will create global unique identifiers and a useful data dictionary as much as we are able in order to deposit data into the National Database allowing other researchers and NIMH to use available data.
  In line with accepted data sharing practices and ethical principles, we will share de-identified raw data with other researchers attempting to replicate our findings or including our findings in subsequent projects.
Supporting Information: Study Protocol
Time Frame: One year after the final results have been published.
Access Criteria: Researchers will be able to contact us by telephone or email to request these data, which we will provide in a timely manner. We will not release any data that are considered identifying or protected by IRB, HIPAA, or federal regulations unless that researcher and the PI of the current project have obtained proper administrative agreements or participation in the NIMH national database.

REFERENCES:
- [Derived] Levin JB, DelBello M, Modi AC, Briggs F, Forthun LF, McVoy M, Yala J, Cooley R, Black J, Conroy C, Sajatovic M. A 6-month, prospective, randomized controlled trial of customized adherence enhancement versus a bipolar-specific educational control in poorly adherent adolescents and young adults living with bipolar disorder. Bipolar Disord. 2024 Nov;26(7):696-707. doi: 10.1111/bdi.13489. Epub 2024 Sep 4. PMID 39231780

RESULTS

PARTICIPANT FLOW:
Period: Baseline (Randomized)
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0
Period: Week 8
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
Started | 17 | 19
Completed | 15 | 15
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Suspended | 0 | 1
Period: Week 12
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: Week 24
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
Started | 13 | 13
Completed | 11 | 12
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU) | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.2 (2.3) | 19.1 (1.8) | 19.1 (2.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 2 | 6 | 8
  Gender: Female | 13 | 11 | 24
  Gender: Other | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 13 | 15 | 28
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Age diagnosed with Bipolar Disorder [Mean (Standard Deviation); unit: years] | 15.7 (4.8) | 16.3 (3.6) | 16 (4.1)
Current living situation [Count of Participants; unit: Participants]
  Living Alone | 4 | 0 | 4
  With parents/guardian/caregiver | 6 | 12 | 18
  Living with others | 7 | 7 | 14
Household income [Count of Participants; unit: Participants]
  0-35K | 6 | 6 | 12
  36-75k | 4 | 3 | 7
  76-150k | 3 | 2 | 5
  150k+ | 1 | 3 | 4
  Decline/Don't Know | 3 | 5 | 8
Years of education [Mean (Standard Deviation); unit: years] | 12.6 (2.2) | 12.8 (1.6) | 12.7 (1.9)
Hospitalization history [Count of Participants; unit: Participants]
  Yes | 11 | 9 | 20
  No | 6 | 10 | 16
Family History of Bipolar Disorder [Count of Participants; unit: Participants]
  Yes | 9 | 14 | 23
  No | 8 | 4 | 12
  Don't Know | 0 | 1 | 1
Attention-deficit/hyperactivity disorder Diagnosis [Count of Participants; unit: Participants]
  Yes | 8 | 14 | 22
  No | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Tablet Routine Questionaire (TRQ) "Past Month" Item at 24 Weeks
Description: The TRQ "past month" item is a subject report of the percentage of prescribed medications not taken within the past month.
Time Frame: Baseline and 24 weeks
Population: Only those with complete data for TRQ past month at baseline and 24 weeks were included in the analysis
Measure: Mean (Standard Deviation); unit: percent of medications not taken
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
Number analyzed (Participants) | 11 | 11
percent of medications not taken | 21.5 (17.0) | 28.0 (35.8)

2. Primary Outcome: Change From Baseline in the Tablet Routine Questionaire (TRQ) "Past Week" Item at 24 Weeks
Description: The TRQ "past week" item is a subject report of the percentage of prescribed medications not taken within the past week.
Time Frame: Baseline and 24 weeks
Population: Only those with complete data for TRQ past week at baseline and 24 weeks were included in the analysis
Measure: Mean (Standard Deviation); unit: percent of medications not taken
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
Number analyzed (Participants) | 11 | 11
percent of medications not taken | 27.9 (27.9) | 28.6 (36.1)

3. Primary Outcome: Change From Baseline in Treatment Adherence as Measured by Special Pill Counter at 24 Weeks
Description: A special pill cap/box will record the time/date of bottle opening. A dose will be counted as "taken" if the bottle is opened within two hours of the prescribed time. A percent of doses taken (treatment adherence) will be calculated by dividing the number of times the bottle is opened by the number of times it should have been opened as per the prescription.
Time Frame: Baseline and 24 weeks
Population: Only those with complete data from the pill counter at baseline and 24 weeks were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of doses taken
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
Number analyzed (Participants) | 4 | 4
percentage of doses taken | 85.7 (16.5) | 50.0 (36.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period of 6 months.
Arm/Group | Customized Adherence Enhancement for AYA | Enhanced Treatment as Usual (ETAU)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Customized Adherence Enhancement for AYA (N=17) | Enhanced Treatment as Usual (ETAU) (N=19)
Hospitalization for Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Hospitalization for Severe Electrolyte Imbalance (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT04348604/Prot_SAP_000.pdf